CLINICAL TRIAL: NCT02514538
Title: EVALUATION OF THE RELATIONSHIP BETWEEN EFFERVESCENT PARACETAMOL AND BLOOD PRESSURE. CLINICAL TRIAL.
Acronym: Paracetamol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IJG-PAR-2010
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension; Chronic Disease of Musculoskeletal System
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-effervescent tablets (Experimental): Comparing the effect of two different formulations of paracetamol (effervescent or non-effervescent tablets) in the blood pressure of hypertensive patients after 3 weeks treatment . The washing time between the two periods is approximately 1 week (minimum 3 days).
  Interventions: Drug: Non- effervescent Paracetamol kern; Drug: Effervescent paracetamol termalgin
- Effervescent Paracetamol (Active Comparator): Comparing the effect of two different formulations of paracetamol (effervescent or non-effervescent tablets) in the blood pressure of hypertensive patients after 3 weeks treatment . The washing time between the two periods is approximately 1 week (minimum 3 days).
  Interventions: Drug: Non- effervescent Paracetamol kern; Drug: Effervescent paracetamol termalgin

INTERVENTIONS:
Drug: Non- effervescent Paracetamol kern — 1g
Drug: Effervescent paracetamol termalgin — 1 g

SUMMARY:
Paracetamol's solubility is achieved by adding to the excipient sodium salts, either as bicarbonate, carbonate or citrate. As the relationship between salt and hypertension is well known, due to the sodium content it has raised a hypothesis that may interfere with the control of that risk factor.

Therefore, the objective of this study is to evaluate the effect on blood pressure of effervescent paracetamol compared to non-effervescent, in hypertensive patients.

This is a multicenter, randomized, controlled, crossover, open, phase IV clinical trial, which compares the effect of two different formulations of paracetamol (effervescent or non-effervescent tablets) in the blood pressure of hypertensive patients after 3 weeks treatment (coded EUDRACT 2010-023485-53). The washing time between the two periods is approximately 1 week (minimum 3 days)

DETAILED DESCRIPTION:
Inclusion criteria:

Patients included in the study must meet the following criteria:

* be hypertensive patients over 18 years
* with degenerative joint disease
* which regularly need analgesic treatment. They must submit BP in the consultation lower than 150 and 95 mmHg or lower than 135 and 85 mmHg if they have associated cardiovascular disease (stroke, coronary heart disease, peripheral arterial disease) or diabetes mellitus.

They can't receive pharmacological antihypertensive treatment, or this must be stable and unchanged in the last month.

In relation to osteoarticular disease, they should have a degree of mild to moderate pain, with a score between 1 and 4 on a visual analog scale (VAS)

Evaluation of results

Primary endpoint:

The primary endpoint is the change in mean daytime, night-time (sleep) and 24-hour systolic BP, measured by ABPM, from baseline at 3 weeks of treatment in both periods.

Secondary endpoints:

* Changes in systolic BP measured in the clinic at the end of 3-week follow-up respect baseline in both periods.
* 24-hour, daytime and night-time (sleep) diastolic BP measured by ABPM: change from baseline at 3 weeks of treatment in both periods
* Changes in diastolic BP measured in the clinic at the end of 3-week follow-up respect baseline in both periods.
* Percentage of patients maintaining clinical BP under 140 and 90 mmHg at the end of each period
* Degree of pain assessed by visual analog scale
* Consumption of rescue medication
* Therapeutic compliance

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study must meet the following criteria:
* be hypertensive patients over 18 years
* with degenerative joint disease
* which regularly need analgesic treatment. They must submit BP in the consultation lower than 150 and 95 mmHg or lower than 135 and 85 mmHg if they have associated cardiovascular disease (stroke, coronary heart disease, peripheral arterial disease) or diabetes mellitus.

They can't receive pharmacological antihypertensive treatment, or this must be stable and unchanged in the last month.

In relation to degenerative joint disease, they should have a degree of mild to moderate pain, with a score between 1 and 4 on a visual analog scale (VAS)

Exclusion Criteria:

* Patients with allergy, intolerance or contraindication to paracetamol or tramadol will be excluded, as those who have taken nonsteroidal antiinflammatory drugs (NSAIDs) orally or parenterally in the last week, or have a high degree of pain (VAS> 4) or poorly controlled hypertension (office BP> 150/95 mmHg or daytime ambulatory mean BP > 140/90 mmHg).

Patients with heart failure due to systolic and / or diastolic dysfunction will also be excluded, those who have suffered a cardiovascular event (myocardial infarction, unstable angina or stroke of any type) in the last 6 months, presenting sleep apnea or any form of secondary hypertension, elevated transaminases (higher than 3 times normal value), or a glomerular filtration rate <30 ml/min, over a maximum period of three months before starting the study; patients with dementia or judicial disability, with alcoholism or other addictions; pregnant patients; patients treated with oral anticoagulants or subcutaneous heparin. Patients in which changes are foreseen in usual dose drugs with effects on BP throughout the study (alpha blockers, tricyclic antidepressants, beta blockers in eye drops, sympathomimetic vasoconstrictor, other effervescent agents, hormonal contraceptives, NSAIDs, corticosteroids, anabolic, erythropoietin, cyclosporine) or those who will initiate major changes in lifestyles (onset or increase physical exercise, dietary changes); those who do not give their informed consent and that in the opinion of the investigator, have poor adherence or may become lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
value of BP measured by ABPM | 3 Weeks
  The primary endpoint is the change in mean daytime, night-time (sleep) and 24-hour systolic BP, measured by ABPM, from baseline at 3 weeks of treatment in both periods.

REFERENCES:
- [Derived] Benitez-Camps M, Vinyoles-Bargallo E, Rebagliato-Nadal O, Morros-Pedros R, Pera-Pujadas H, Dalfo-Baque A, Lopez-Pavon I, Roca-Sanchez C, Coma-Carbo RM, De La Figuera Von Wichmann M, Mengual-Martinez L, Yuste-Marco C, Teixido-Colet M, Pepio i Vilaubi JM, Ciurana-Tost R, Pou-Vila R, Vila-Coll MA, Bordas-Julve JM, Aragones-Fores R, Pelegrina-Rodriguez FJ, Agudo-Ugena J, Blanco-Mata C, de la Iglesia Berrojalbiz J, Burgos-Alonso N, Gomez-Fernandez MC. Evaluation of the relationship between effervescent paracetamol and blood pressure: clinical trial. BMC Cardiovasc Disord. 2015 Dec 10;15:167. doi: 10.1186/s12872-015-0161-7. PMID 26654907